CLINICAL TRIAL: NCT06357182
Title: A Phase Ib Investigation of the LSD1 Inhibitor Iadademstat (ORY-1001) in Combination With Azacitidine and Venetoclax in Newly Diagnosed AML
Brief Title: Iadademstat in Combination With Azacitidine and Venetoclax in Treating Newly Diagnosed Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other); Oryzon Genomics S.A. (Industry)
Responsible Party: Principal Investigator, Curtis Lachowiez, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00026136; NCI-2024-01262 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00026136 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2024-02-29; First posted 2024-04-10 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome/Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; GATA2 Deficiency | interventions — Azacitidine; Specimen Handling; Biopsy; iadademstat; venetoclax

STUDY DESIGN:
Intervention Model Description: The treatment plan starts with a 7 day monotherapy lead-in (Cycle 0 [C0]) and then proceeds to combination therapy in 28 day cycles. Disease will be assessed pre-treatment (Screening/Baseline), at the end of monotherapy, in C1 (and C2, if response is not observed in C1), and at the end of alternating cycles, thereafter. A disease assessment will also be conducted within 30 days of the last dose of IADA. Participants that do not achieve response after up to 2 cycles of the triplet regimen will be taken off treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment Dose Level -1 (iadademstat, azacitidine, venetoclax) (Experimental): Iadademstat (75 mcg, 5+2 days, 2 out of 4 weeks per cycle), Venetoclax (400 mg, day 1-14), Azacitidine (75 mg/m2, day 1-7)
  Patients receive iadademstat PO QD on days 1-5 of cycle 0 and then days 1-5, 8-12, and 15-19. Patients also receive venetoclax PO QD days 1-21 and azacitidine SC QD days 1-7. Patients with CR, CRh, CRi, or MLFS after cycle 1 continue to receive IADA PO QD on days 1-5, 8-12, and 15-19, azacitidine SC QD days 1-7 and venetoclax PO QD days 1-21 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO or MUGA during screening as clinically indicated on study. Patients under bone marrow biopsy throughout the trial. Additionally, patients undergo blood sample collection during screening and on the trial.
  Interventions: Drug: Azacitidine; Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Procedure: Echocardiography Test; Drug: Iadademstat; Procedure: Multigated Acquisition Scan; Other: Questionnaire Administration; Drug: Venetoclax
- Treatment Dose Level -2 (iadademstat, azacitidine, venetoclax) (Experimental): Iadademstat (75 mcg, 5+2 days, 2 out of 4 weeks per cycle), Venetoclax (400 mg, day 1-7), Azacitidine (50 mg/m2, day 1-7).
  Patients receive iadademstat PO QD on days 1-5 of cycle 0 and then days 1-5, 8-12, and 15-19. Patients also receive venetoclax PO QD days 1-21 azacitidine SC QD days 1-7. Patients with CR, CRh, CRi, or MLFS after cycle 1 continue to receive IADA PO QD on days 1-5, 8-12, and 15-19, azacitidine SC QD days 1-7 and venetoclax PO QD days 1-21 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO or MUGA during screening as clinically indicated on study. Patients under bone marrow biopsy throughout the trial. Additionally, patients undergo blood sample collection during screening and on the trial.
  Interventions: Drug: Azacitidine; Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Procedure: Echocardiography Test; Drug: Iadademstat; Procedure: Multigated Acquisition Scan; Other: Questionnaire Administration; Drug: Venetoclax
- Treatment Dose Level 1 (iadademstat, azacitidine, venetoclax) (Experimental): Iadademstat (100 mcg, 5+2 days, 2 out of 4 weeks per cycle), Venetoclax (400 mg, day 1-21), Azacitidine (75 mg/m2, day 1-7)
  Patients receive iadademstat PO QD on days 1-5 of cycle 0 and then days 1-5, 8-12, and 15-19. Patients also receive venetoclax PO QD days 1-21 and azacitidine SC QD days 1-7. Patients with CR, CRh, CRi, or MLFS after cycle 1 continue to receive IADA PO QD on days 1-5, 8-12, and 15-19, azacitidine SC QD days 1-7 and venetoclax PO QD days 1-21 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO or MUGA during screening as clinically indicated on study. Patients under bone marrow biopsy throughout the trial. Additionally, patients undergo blood sample collection during screening and on the trial.
  Interventions: Drug: Azacitidine; Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Procedure: Echocardiography Test; Drug: Iadademstat; Procedure: Multigated Acquisition Scan; Other: Questionnaire Administration; Drug: Venetoclax
- Treatment Dose Level 2 (iadademstat, azacitidine, venetoclax) (Experimental): Iadademstat (150 mcg, 5+2 days, 2 out of 4 weeks per cycle), Venetoclax (400 mg, day 1-21), Azacitidine (75 mg/m2, day 1-7)
  Patients receive iadademstat PO QD on days 1-5 of cycle 0 and then days 1-5, 8-12, and 15-19. Patients also receive venetoclax PO QD days 1-21 and azacitidine SC QD days 1-7. Patients with CR, CRh, CRi, or MLFS after cycle 1 continue to receive IADA PO QD on days 1-5, 8-12, and 15-19, azacitidine SC QD days 1-7 and venetoclax PO QD days 1-21 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO or MUGA during screening as clinically indicated on study. Patients under bone marrow biopsy throughout the trial. Additionally, patients undergo blood sample collection during screening and on the trial.
  Interventions: Drug: Azacitidine; Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Procedure: Echocardiography Test; Drug: Iadademstat; Procedure: Multigated Acquisition Scan; Other: Questionnaire Administration; Drug: Venetoclax

INTERVENTIONS:
Drug: Azacitidine — Given SC
  Other Names: 5 AZC; 5-AC; 5-Azacitidine; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Drug: Iadademstat — Given PO
  Other Names: ORY 1001; ORY-1001; RG 6016; RG6016; RO 7051790; RO7051790; trans-N1-((1R,2S)-2-Phenylcyclopropyl)-1,4-cyclohexanediamine
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Other: Questionnaire Administration — Ancillary study
Drug: Venetoclax — Given PO
  Other Names: ABT 199; ABT-0199; ABT-199; ABT199; GDC 0199; GDC-0199; GDC0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of iadademstat when given together with azacitidine and venetoclax in treating patients with newly diagnosed acute myeloid leukemia (AML). Iadademstat inhibits the LSD1 protein and may lead to inhibition of cell growth in LSD1-overexpressing cancer cells. Chemotherapy drugs, such as azacitidine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Venetoclax is in a class of medications called B-cell lymphoma-2 (Bcl-2) inhibitors. It may stop the growth of cancer cells by blocking Bcl-2, a protein needed for cancer cell survival. Giving iadademstat with azacitidine and venetoclax may be safe, tolerable and/or effective in treating patients with newly diagnosed AML who cannot undergo intensive chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D) of iadademstat (IADA) when administered as part of the investigational combination (i.e., iadademstat + azacitidine + venetoclax [IADA+AZA+VEN]).

SECONDARY OBJECTIVES:

I. Assess the preliminary efficacy of the investigational regimen based on disease remission.

II. Assess the preliminary efficacy of the investigational regimen based on clinical response.

III. Assess the safety of the investigational regimen.

EXPLORATORY OBJECTIVES:

I. Assess survival in the absence of treatment failure, hematologic relapse, or progressive disease.

II. Assess overall survival.

III. Assess duration of response, based on morphological assessments.

IV. Identify mechanisms of transcriptional reprogramming and cell death.

V. Identify predictive biomarkers of response to LSD1 inhibition.

VI. Assess participant quality of life using Patient-Reported Outcomes Common Terminology Criteria for Adverse Events (PRO-CTCAE).

OUTLINE: This is a dose-escalation study of iadademstat in combination with azacitidine and venetoclax.

Patients receive iadademstat orally (PO) once daily (QD) on days 1-5, 8-12, and 15-19. Patients also receive venetoclax PO QD days 1-21 or 1-28 and azacitidine subcutaneously (SC) QD days 1-7. Patients with complete remission (CR), CR with partial hematologic recovery (CRh), CR with incomplete blood count recovery, (CRi), or morphologic leukemia-free state (MLFS) after cycle 1 continue to receive IADA PO QD on days 1-5, 8-12, and 15-19, azacitidine SC QD days 1-7 and venetoclax PO QD days 1-21 or 1-28 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients undergo echocardiography (ECHO) or multigated acquisition scan (MUGA) during screening as clinically indicated on study. Patients under bone marrow biopsy throughout the trial. Additionally, patients undergo blood sample collection during screening and on the trial.

After completion of study treatment, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years of age will be considered for inclusion without bias against gender identity, race, or ethnicity
* Ability to comprehend the investigational nature of the study and provide written informed consent
* Patients with previously untreated, morphologically documented AML based on World Health Organization (WHO) 2008 definitions who are ineligible for standard of care (SOC) intensive chemotherapy induction and also meet the following criteria:

  * Documented intermediate- or adverse-risk AML based on European Leukemia Network (ELN) 2022 criteria
  * Note: Cases of AML/myelodysplastic syndrome (MDS) overlap with 10-19% bone marrow (BM) or peripheral blood (PB) blasts will be considered
  * Note: Cases of acute promyelocytic leukemia (PML) and AML with BCR::ABL1 fusions will be excluded
* Eastern Cooperative Oncology Group (ECOG) performance ≤ 2 (Patients aged ≥ 75 years, at the time of consent)
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN) (Patients aged ≥ 75 years, at the time of consent)

  * High total bilirubin values may require indirect and direct bilirubin testing. Individuals with known Gilbert's syndrome may be considered for enrollment despite high indirect (and total) bilirubin
* Creatinine clearance (CrCl) of ≥ 60 mL/min (estimated using the Cockcroft Gault formula or measured by 24 hours urine collection. If altered, CrCl is determined to be related to concomitant medication that alters renal function
* Patients aged ≥ 18 to 74 years (ECOG performance status [PS] ≤ 3 is accepted) at consent must meet ≥ 1 of the following criteria defining a co morbidity:

  * ECOG PS of 2 or 3 (Note: Patients ≥ 18 to 74 years of age with PS of 0-1 must meet criteria of one of the following comorbidities.)
  * Cardiac history of congestive heart failure (CHF) requiring treatment or ejection fraction ≤ 50% or chronic stable angina
  * Diffusing capacity of the lung for carbon monoxide (DLCO) ≤ 65% or forced expiratory volume in 1 second (FEV1) ≤ 65%
  * CrCl ≥ 30 mL/min to < 45 ml/min
  * Moderate hepatic impairment with total bilirubin > 1.5 to ≤ 3.0 × ULN;

    * High total bilirubin values may require indirect and direct bilirubin testing. Individuals with known Gilbert's syndrome may be considered for enrollment despite high indirect (and total) bilirubin
  * Other comorbidities that the physician judges to be incompatible with intensive chemotherapy (IC). In these cases, the comorbidity must be reviewed and approved by the principal investigator (PI) before study enrollment
* Ability to swallow oral medications
* No ongoing anticoagulation or antiplatelet therapy within 14 days of start of treatment with IADA
* No history of severe bleeding disorder such as hemophilia A, hemophilia B, von Willebrand disease, or history of spontaneous bleeding requiring blood transfusion or other medical intervention
* No history of stroke or intracranial hemorrhage within 180 days of start of IADA
* No major bleeding event, as defined by the International Society of Thrombosis and Hemostasis (ISTH), within 12 weeks of start of IADA
* Uncorrected international normalized ratio (INR) or activated partial thromboplastin time (aPTT) of < 1.5 x ULN.

  * If INR or aPTT > 1.5 x ULN has been corrected (prior to enrollment), then history of disseminated intravascular coagulation (DIC) must be absent
* White blood cell (WBC) < 20 x 10^9/L prior to study start. Cytoreduction prior to study treatment is allowed with

  * Hydroxyurea for up to 14 days and until 24 hours prior to start of IADA; or
  * Leukapheresis for up to 14 days prior to start of IADA
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) or alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) ≤ 2.0 x institutional ULN

  * Lower hepatic function may be considered if liver enzyme abnormalities are determined by the treating MD and principal investigator (PI) to be due to leukemic infiltration
* Willing and able to

  * Adhere to study schedule of activities and life style restrictions while on treatment;
  * Provide bone marrow (BM) aspirate and core biopsy samples; and
  * Accept supportive and prophylactic care for hematologic toxicities, infection, and immediate sequelae, including transfusions
* Negative pregnancy test within 72 hours of start of IADA for persons of childbearing potential (PCBP)
* Willingness to comply with study requirements for contraception, as follows: PCBP and sperm-producing participants who are sexually active with a PCBP must use study approved contraception from start of investigational product (first dose of IADA) until 6 months after the last dose of IADA. Pregnancy is exclusionary because the agents used in this study have the potential for teratogenic or abortifacient effects

Exclusion Criteria:

* Prior allergic response to iadademstat (IADA), venetoclax, azacitidine, or any excipients in the formulations
* Body weight < 50 kg
* Investigational therapy within 5 half-lives or, if unknown, within 28 days prior to start of IADA
* Treatment for AML within 14 days prior to start of IADA. Cytoreduction for patients with proliferative disease must meet the criteria listed in inclusion criteria
* Radiotherapy less than 14 days prior to start of IADA
* Recent and significant medical interventions, such as major surgery within 28 days prior to the start of IADA, or stem cell transplant within 100 days prior to the start of IADA. Patients with active treatment for graft-versus-host disease (GVHD) are excluded
* Another active malignancy within 5 years prior to the start of IADA, or at the investigator's discretion
* Treatments targeting or inhibiting LSD1/KDM1A or BCL 2 within 12 months prior to the start of IADA
* Documented dysphagia, short-gut syndrome, gastroparesis, or other conditions that limit the ingestion or gastrointestinal absorption of drugs administered orally
* Treatment with monoamine oxidase inhibitors (e.g., tranylcypromine), if treatment is not finalized at least 3 weeks prior to the start of IADA
* Active central nervous system involvement with AML
* Uncontrolled infection. Participants with controlled infection must be afebrile and hemodynamically stable for at least 72 hours prior to start of IADA and must be amenable to alternate treatment if current treatment will interact with investigational regimen
* Active hepatic disorder or documented positive hepatitis B or C virus (HBV/HCV, respectively) status, except in cases of undetectable HBV/HCV viral load for at least 3 months prior to the start of IADA. (Hepatitis B or C testing is not required for eligibility assessment.)
* Individuals serology positive for human immunodeficiency virus (HIV) and under active treatment with highly active antiretroviral therapy (HAART) (or another therapy that may interfere with metabolism of study agents). Otherwise, enrollment may be considered in cases of HIV that is controlled with another treatment type or in cases that that acceptable modification of the patient's HIV treatment exists
* Use a P-gp inhibitor within 21 days or 3 half-lives whichever is longer prior to treatment with venetoclax
* Use of strong or moderate CYP3A4 inducers or inhibitors within 2 days or 3 half lives whichever is longer, prior to start of treatment with venetoclax
* Unwillingness to stop breastfeeding. Because there is a potential risk for adverse events in nursing infants secondary to treatment of the mother with the chemotherapy agents, breastfeeding should also be avoided throughout the study and until at least 60 days after last dose of IADA
* Uncontrolled hypertension (i.e., systolic blood pressure > 180 mm Hg, diastolic blood pressure > 95 mm Hg). Use of anti-hypertensive agents to control hypertension before C1D1 is allowed
* Patients with poorly controlled diabetes. Poorly controlled diabetes mellitus defined as glycosylated hemoglobin (HbA1c) ≥ 8%; patients with a history of transient glucose intolerance due to corticosteroid administration may be enrolled in this study if all other inclusion/exclusion criteria are met
* Patients with mean of triplicate corrected QT interval (Fridericia's correction formula [QTcF]) > 450 ms at Screening based on central reading
* Uncontrolled intercurrent illness including, but not limited to ongoing or active uncontrolled infection, unstable cardiac or pulmonary function or acute insufficiency (e.g., symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia), or psychiatric illness or social situation that could limit compliance with study requirements, at the discretion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-08-22 (Actual); Primary Completion 2026-03-08 (Estimated); Study Completion 2026-05-29 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) within specific iadademstat (IADA) dose levels | Start of IADA (cycle 1 of combination therapy) to end of cycle 1 (each cycle is 28 days)
  Will be assessed by National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v 5.0).

SECONDARY OUTCOMES:
Percentage of efficacy-evaluable participants achieving composite complete remission (cCR) | Start of IADA (cycle 1 of combination therapy) to end of investigational study treatment, average of 1 year
  Will be defined as achievement of complete remission (CR) or CR with partial hematologic recovery (CRh) or CR with incomplete blood count recovery (CRi) while on iadademstat+ azacitidine + venetoclax (IADA+AZA+VEN). Will be estimated for the efficacy-evaluable population with point estimates and exact binomial confidence intervals (CIs) as summary statistics. CRc rate will also be modeled with univariable logistic regressions to determine if any baseline patient or disease feature is correlated with clinical response as defined by these efficacy metrics.
Percentage of efficacy-evaluable participants achieving an overall response (ORR) | Start of IADA (cycle 1 of combination therapy) to end of investigational study treatment, average of 1 year
  Will be defined as the proportion of efficacy-evaluable participants who attain a PR or better (i.e., CR, CRh, CRi, morphologic leukemia-free state, or partial remission [PR]) while on IADA+AZA+VEN. Will be estimated for the efficacy-evaluable population with point estimates and exact binomial CIs as summary statistics. ORR will also be modeled with univariable logistic regressions to determine if any baseline patient or disease feature is correlated with clinical response as defined by these efficacy metrics.
Incidence of treatment-emergent grade ≥ 3 adverse events (AEs) | Start of IADA (cycle 1 of combination therapy) to end of investigational study treatment, average of 1 year
  Will be reported with descriptive statistics, at the overall patient level and by grade, attribution (i.e., a separate table for treatment-related AEs), and seriousness (i.e., separate tables for serious adverse events).

CONTACTS AND LOCATIONS:
Overall Officials: Curtis A Lachowiez, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States